CLINICAL TRIAL: NCT05623644
Title: Multimodal MR Imaging Study on ET and PD Patients Subjected With MRgFUS Thalamotomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Chairman of the Department of Radiology, Chinese PLA General Hospital
Other Study IDs: MRgFUS-VIM-prospective-2022
Record Dates: First submitted 2022-11-12; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Movement Disorders
Keywords: Essential tremor; Parkinson disease; MRgFUS; Magnetic resonance imaging
MeSH Terms: conditions — Movement Disorders; Essential Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TD-PD patients undergoing MRgFUS thalamotomy: The imaging data from patients with tremor dominant PD underwent MRgFUS thalamotomy. Their clinical and imaging data were also collected.
- MR-ET patients undergoing MRgFUS thalamotomy: The imaging data from patients with medication-resistant ET underwent MRgFUS thalamotomy. Their clinical and imaging data were also collected.

SUMMARY:
The technological advance of magnetic resonance-guided focused ultrasound (MRgFUS) has once again brought lesion therapy back to the clinical frontline for the treatment of movement disorder. Thus far, the safety of MRgFUS has been widely proven and has just been made available in China in late 2020. We attempted to analyze the neuroplasticity characteristics and altered neural circuit activity in patients subjected with MRgFUS thalamotomy via Multiple MR Imaging study, and to explore potential biomarkers that could be used to predict the treatment outcome.

DETAILED DESCRIPTION:
Essential tremor (ET) and Parkinson disease (PD) are the most prevalent tremor disorders. ET, considered as a pure tremor disease, is characterized by upper limb intention or postural tremor, while PD is characterized by a variety of motor and nonmotor symptoms, among them rest tremor. Tremor suppression can be achieved by lesioning or stimulating a relay nucleus of the thalamus, known as the ventral intermediate nucleus (VIM). One emerging and promising approach to lesion VIM is magnetic resonance-guided focused ultrasound (MRgFUS). This technique allows delivery of spherical phased converging beams to a specific brain target using MR imaging (MRI) for guidance. A number of studies have demonstrated the effectiveness and safety of ExAblate MRgFUS thalamotomy for medication-refractory tremor in patients with ET/PD. MRgFUS thalamotomy has been approved for ET/PD patients in late 2020.

Magnetic resonance imaging (MRI) is a technique for measuring structural features and mapping brain activity that is noninvasive and safe. It is being used in many studies to better understand how the healthy brain works, and in a growing number of studies it is being applied to understand how that normal function is disrupted in disease. The analysis of the imaging data related to MRgFUS thalamotomy may help us to further understand the neuroplasticity characteristics of patients around treatment and the altered brain network dynamics. It would also further help us grasp the advantages and disadvantages of such brain lesion therapy techniques and serves guidance for the next clinical studies. Therefore, we registered this new study for our current prospective study.

Brief summary of retrospective data：

- Medication-refractory ET and PD Patients subjected with MRgFUS thalamotomy were recruited for multimodal MR scanning, including T2; T2 Flair; DWI; ESWAN; MRS; 3D ASL 2.0s; 3D-T1; DTI; rs-functional MRI at baseline, postoperative 1-day, postoperative 1-week, postoperative 1-month, postoperative 3-months, postoperative 6-months, postoperative 1-year, postoperative 2-year, postoperative 3-year, postoperative 4-year, postoperative 5-year. Extra baseline info were also collected, as well as ultrasound parameters (energy, power, duration time, temperature, target location), clinical assessment (clinical rating scale for tremor (CRST), Unified Parkinson Disease Rating Scale (UPDRS), associated adverse effects and so on.

ELIGIBILITY:
* Inclusion Criteria:

  1. Any patient who intends to undergo MRgFUS thalamotomy for tremor control will be recruited for additional multimodal MR Imaging scranning；
  2. A clear diagnosis of ET and PD as confirmed from clinical history and examination by a neurologist or neurosurgeon specialized in movement disorder;
  3. Men and women age 18 years or older;
  4. Intolerance to side effects of medication or poor response to medication, severe and disabling tremor;
  5. Able to communicate sensations during the ExAblate TcMRgFUS treatment;
  6. Having complete medical history and clinical follow up;
  7. MR Imaging scanning can be processed.
* Exclusion Criteria:

  1. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc;
  2. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease;
  3. Subjects with unstable cardiac status;
  4. Severe hypertension (diastolic BP > 100 on medication);
  5. Patient with severely impaired renal function;
  6. History of abnormal bleeding and/or coagulopathy;
  7. History of immunocompromise including those who are HIV positive;
  8. History of intracranial hemorrhage;
  9. Cerebrovascular disease (multiple CVA or CVA within 6 months);
  10. Subjects with uncontrolled symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, papilledema);
  11. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time);
  12. Significant claustrophobia that cannot be managed with mild medication;
  13. Presence of any other neurodegenerative disease such as Parkinson-plus syndromes suspected on neurological examination;
  14. Presence of significant cognitive impairment;
  15. Subjects with life-threatening systemic disease;
  16. Subjects with a history of seizures within the past year;
  17. Subjects with presence or history of psychosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ET and PD patients subject with MRgFUS thalamotomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Tremor measurement in ET/PD patients subject with MRgFUS thalamotomy | 5 years
  The change in the hand tremor score derived by summing eight items of the CRST/UPDRS that evaluate hand tremor and ability to perform tasks will be evaluated for movement disorders subjects.
Adverse reactions in ET/PD patients subject with MRgFUS thalamotomy | 5 years
  Adverse Events will be evaluated using Significant Clinical Complications for movement disorders subjects. Adverse Events will be reported and categorized by investigators as definitely, probably, possibly, or unrelated to the device or procedure and categorized by treatment group / treatment arm.
Imaging features in ET/PD patients subject with MRgFUS thalamotomy | 5 years
  Lesion appearance and volume are measured by T2, T2 Flair, DWI, ESWAN, 3D-T1; ESWAN and MRS manifests the changes of iron deposition and metabolism, respectively; ASL shows regional cerebral blood flow associated with the procedure; DTI demonstrates the destruction of white matter integrity and structural network; Rs-functional MRI reflects alterations of resting-state brain activity and functional network; others.
Postoperative symptom recurrence of patients Postoperative symptom recurrence of patients Postoperative symptom recurrence of patients Postoperative symptom recurrence of patients Postoperative symptom recurrence of patients | 5 years
  It has been reported in the previous literature that about 10%-50% of the patients with MRgFUS thalamotomy had recurrent symptoms after the operation. We mainly recorded the recurrence of tremor in patients and the clinical symptoms and signs associated with this process in a long-term longitudinal observation.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD/PhD, Principal Investigator — Chinese PLA General Hospital; LongSheng Pan, MD/PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Jiaji Lin, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided